CLINICAL TRIAL: NCT00988910
Title: Observational Study on the Effects of DRSP-Containing Combined Oral Contraceptives (Yasmin,Yasminelle) and Other Combined Oral Contraceptives on the General and Sexual Well-Being in COC Users
Brief Title: Effects of Drospirenone-containing or -Not Containing Combined Oral Contraceptives on General and Sexual Well-being
Acronym: COSME
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14182; YA0711IT (Other: Other company ID)
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Contraception
Keywords: Combined Oral Contraceptives; COC
MeSH Terms: interventions — drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1
  Interventions: Drug: EE30-DRSP (Yasmin, BAY86-5131)
- Group 2
  Interventions: Drug: Other combined oral contraceptives

INTERVENTIONS:
Drug: EE30-DRSP (Yasmin, BAY86-5131) — DRSP-containing combined oral contraceptives according to the normal routine praxis
  Groups: Group 1
Drug: Other combined oral contraceptives — Other combined oral contraceptives according to the normal routine praxis
  Groups: Group 2

SUMMARY:
The purpose of this study is to evaluate the symptoms and satisfaction for women taking drospirenone (DRSP)-containing combined oral contraceptives in comparison with women taking other kind of combined oral contraceptives.

ELIGIBILITY:
Inclusion Criteria:

* According to the label of the prescribed Combined Oral Contraceptive (COC)
* first Combined Oral Contraceptive use or previous Combined Oral Contraceptive use
* intention to use current COC for 1 year at least

Exclusion Criteria:

* Contraindications listed in the label of the prescribed Combined Oral Contraceptive (COC)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women using Combined Oral Contraceptive (COC)
Sampling Method: Non-Probability Sample
Enrollment: 632 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Psychophysical well-being evaluated by the Psychological General Well-Being Index (PGWBI) | at 12 months
Sexual well-being evaluated by the Female Sexual Function Index (FSFI) | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Italy